CLINICAL TRIAL: NCT00690352
Title: Comparing Recidivism Rates of Felony Drug Offenders in Nebraska Who Were Sentenced to, and/or Participated in, Specialized Substance Abuse Supervision (SSAS) to Those Without SSAS
Brief Title: Specialized Substance Abuse Supervision (SSAS) Versus Non-SSAS Recidivism Rates Among Nebraska Felony Drug Offenders
Acronym: SSAS
Status: Completed | Type: Observational
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Other Study IDs: 0066-08-FB
Record Dates: First submitted 2008-05-06; First posted 2008-06-04 (Estimated); Last update posted 2023-09-25 (Actual); Status verified 2023-09

CONDITIONS: Substance-related Disorders; Alcohol-related Disorders
Keywords: Specialized Substance Abuse Supervision; SSAS; substance use disorder; felony drug offender; probation; parole; cognitive behavioral therapy; CBT
MeSH Terms: conditions — Substance-Related Disorders; Alcohol-Related Disorders | interventions — Motivational Interviewing

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Specialized Substance Abuse Supervision (SSAS) — Six months participation in SSAS which may include cognitive behavioral therapy (CBT) in groups; use of incentives, positive reinforcement, and/or motivational interviewing.
  Other Names: CBT; motivational interviewing; positive reinforcement; use of incentives

SUMMARY:
This social science study hypothesizes that convicted felony drug offenders in Nebraska who participated in Specialized Substance Abuse Supervision (SSAS) as part of their probation or parole showed significantly better outcomes (specifically, less recidivism) at six months post-entrance to SSAS compared to those who did not participate in SSAS.

DETAILED DESCRIPTION:
Since March 2006, Specialized Substance Abuse Supervision (SSAS) has been available at five sites in Nebraska as an enhancement of probation and parole for felony drug offenders whose scores on initial screening instruments warrant such placement. SSAS enhancements to traditional probation and parole include cognitive behavioral therapy (CBT) in groups; use of incentives; positive reinforcement; and motivational interviewing.

Records of probationers and parolees who participated in SSAS starting anytime between March 1, 2006 and February 28, 2007 were studied to assess recidivism rates. Recidivism for this study is defined as "an arrest and conviction on a new charge while on probation or parole."

The records of a matched control group of non-SSAS probationers and parolees who entered probation or parole during the same time period with similar drug felony offenses and similar screening scores were also studied. Control group was also matched, as much as possible, with similar age group, demographic data, rural/urban residence, and level of felony offense.

Investigators performed a statistical analysis to determine recidivism rates at six months post-entrance to SSAS (and for the control group, at six months post-entrance to probation or parole).

ELIGIBILITY:
Inclusion Criteria:

* convicted felony drug offender
* sentenced in Nebraska
* probationer or parolee
* entered probation or parole or SSAS between March 1, 2006 and February 28, 2007

Exclusion Criteria:

* convicted felony drug offender sentenced in Nebraska starting probation or parole between March 1, 2006 and February 28, 2007 who does not match SSAS probationers/parolees in terms of age, demographics, urban v. rural residence, and/or class of felony drug offense.

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Probationers and parolees who participated in SSAS starting anytime between March 1, 2006 and February 28, 2007 at any of the five participating SSAS sites in Nebraska, plus matched sets of probationers and parolees who did not participated in SSAS at any of the probation/parole sites in the state of Nebraska.
Sampling Method: Non-Probability Sample
Enrollment: 344 (Actual)
Dates: Start 2008-03-05 (Actual); Primary Completion 2008-07-06 (Actual); Study Completion 2008-08-20 (Actual)

PRIMARY OUTCOMES:
Recidivism | 6 months
  Proportion of individuals who re-offend during the six months following sentencing

SECONDARY OUTCOMES:
Probation Violation | 6 months
  Percentage of individuals who violated probation during the six months following sentencing
Probation violation with incarceration | 6 months
  Percentage of individuals who violated probation and were incarcerated during the six months following sentencing
Positive drug screens | 6 months
  Percentage of individuals with positive drug screens during the six months following sentencing
Employed | 6 months
  Percentage of individuals employed during the six months following sentencing

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen M Grant, MD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States